CLINICAL TRIAL: NCT00701753
Title: A Pharmacogenetic Investigation of Antipsychotics in Schizophrenia and Schizophrenia-Like Psychoses
Status: Terminated | Type: Observational
Why Stopped: Insufficient subject recruitment.
Sponsor: TheraGenetics Limited (Industry)
Responsible Party: Dr Janet Munro, TheraGenetics Ltd
Other Study IDs: TheraGenetics-002
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Pharmacogenetic; DNA; RNA; Antipsychotic; Olanzapine; Risperidone; Quetiapine; Personalized medicine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Whole blood DNA RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Olanzapine: Subjects treated with olanzapine as part of their routine clinical care
- Risperidone: Subjects treated with risperidone as part of their routine clinical care
- Quetiapine: Subjects treated with quetiapine as part of their routine clinical care

SUMMARY:
An individual's genetic make-up is known to determine their response to antipsychotic medication. Genetic markers that determine efficacy and side effects of medication may be identified and used to predict treatment outcome.

The study is a naturalistic study of routinely prescribed antipsychotics using outcome measures undertaken as part of the routine clinical care of the cohort. These clinical data are linked with genetic information obtained from DNA and RNA from blood samples undertaken as part of the study.

No alteration is made to the subjects treatment regime or medication.

The study is a two stage investigation:

* The first stage involves the collection of a databank of clinical information and blood samples for DNA and RNA extraction from patients treated with antipsychotic medication.
* The second stage is a molecular genetic investigation of treatment-related genetic factors that may contribute to response prediction and predisposition to side effects.

From these genetic studies pharmacogenetic prediction tests will be validated and/or developed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained
* DSM-IV diagnosis must be one of:

  * schizophrenia
  * schizophreniform
  * schizoaffective
  * delusional disorder
  * brief reactive psychosis
  * psychosis not otherwise specified
* Ethnic origin of both parents must be known
* A minimum of 6 weeks continuous treatment completed with the given antipsychotic, prescribed at least at minimum recommended doses
* Prospectively collected outcome data available (pre-treatment and after at least 6 weeks on treatment)

Exclusion criteria:

* Significant psychiatric or medical co-morbidity including history of:

  * head injury with loss of consciousness
  * seizures
  * neurological disorder
  * mental retardation (DSM-IV)
  * drug or alcohol dependence (DSM-IV)
  * serious physical illness e.g. malignancy, hepatic/renal insufficiency
* Concomitant psychotropic medication that may influence ratings
* Concomitant antipsychotics, antidepressants or mood stabilisers prescribed for >2 weeks during the antipsychotic treatment period rated

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Vancouver Coastal Health
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soma Ganesan, MD, Principal Investigator — Vancouver Coastal Health; Janet Munro, MB BS, Study Director — TheraGenetics Limited
Locations (1):
- Vancouver Coastal Health, Vancouver, British Columbia, Canada